CLINICAL TRIAL: NCT03419052
Title: MIND Food and Speed of Processing Training in Older Adults With Low Education, The MINDSpeed Alzheimer's Disease Prevention Pilot Trial
Brief Title: MINDSpeed Food and Brain Training RCT
Acronym: MINDSpeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Clark, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1703766063; R01AG052439 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Low Education; Cognition; Cognitive Training; Polyphenols
Keywords: randomized controlled trial; cognition; cognitive training; MIND diet; quality of life; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MINDSpeed Intervention (Experimental): Consumption of foods high in polyphenols (i.e., MIND foods) AND speed of processing training
  Interventions: Behavioral: Speed of processing training; Behavioral: MIND foods
- MIND food and training control (Active Comparator): Consumption of foods high in polyphenols (i.e., MIND foods) AND online (inert) games
  Interventions: Behavioral: MIND foods; Behavioral: Cognitive training control
- Control foods and speed of processing training (Active Comparator): Consumption of low polyphenol foods AND speed of processing training
  Interventions: Behavioral: Speed of processing training; Behavioral: Control foods
- Double Control (Sham Comparator): Consumption of low polyphenol foods AND online (inert) games
  Interventions: Behavioral: Cognitive training control; Behavioral: Control foods

INTERVENTIONS:
Behavioral: Speed of processing training — Speed of processing training is provided by the Internet-based BrainHQ program from Posit Science, Inc. BrainHQ contains five different speed training modules (Hawk Eye, Visual Sweeps, Fine Tuning, Eye for Detail, Sound Sweeps) which tap time-order judgment, visual discrimination, spatial-match, forward-span, instruction-following, and memory.
  Arms: Control foods and speed of processing training; MINDSpeed Intervention
Behavioral: MIND foods — The "MIND" diet (created by the Rush Aging & Memory group) specifically emphasizes foods high in polyphenols such as berries, nuts, cocoa, black beans, olive oil, and green leafy vegetables. Participants select these foods from the digital study application and receive them through home delivery.
  Arms: MIND food and training control; MINDSpeed Intervention
Behavioral: Cognitive training control — Control training is provided by the Internet-based BrainHQ program from Posit Science, Inc.These are inert games such as tic-tac-toe, connect 4, battleship, etc.
  Arms: Double Control; MIND food and training control
Behavioral: Control foods — Foods contain low polyphenols. Participants select these foods from the digital study application and receive them through home delivery.
  Arms: Control foods and speed of processing training; Double Control

SUMMARY:
The purpose of this study is to learn how foods high in polyphenols and brain training exercises affect older adults' cognitive performance

DETAILED DESCRIPTION:
Adults with low education who give informed consent will complete a baseline cognitive assessment and then be randomized to one of four arms: 1) MIND foods and cognitive training, 2) MIND foods and control training, 3) control foods and cognitive training, or 4) control foods and control training.

All interventions are conducted through applications running on a tablet computer device that we will provide to all participants for the study duration. Cognitive training is delivered through the online BrainHQ program from Posit Science, Inc. The foods will be shown on the tablet device in an online shopping format. Selected foods will be prepared and delivered by the study team.

Active intervention will last for 12 weeks. After the 12-weeks, free food deliveries will cease but participants who were allocated to cognitive training will continue to have access to BrainHQ. Those in the MIND food arms will be encouraged to maintain MIND food consumption.

ELIGIBILITY:
Inclusion criteria:

* age 60 years or older,
* ≤ 12 years of education,
* English speaking,
* Marion County (and immediately surrounding counties) resident, with steady/fixed residence to receive food deliveries
* natural-born US citizen.

Exclusion criteria:

* living in nursing home
* self-reported diagnosis of dementia, Alzheimer's disease (AD), cancer with short life expectancy, multiple sclerosis, epilepsy, schizophrenia, bipolar disorder, Parkinson disease; current chemotherapy or radiation therapy; history of brain tumor, brain surgery, brain infection; stroke or myocardial infarction within the past 12 months
* current alcohol consumption ≥8 drinks per week for women or ≥15 drinks per week for men;
* poor vision (self-reported difficulty reading a newspaper) or color blind;
* low communicative ability (examiner rated) that would interfere with interventions and assessments;
* prior involvement in similar cognitive training studies;
* unable or unwilling to provide blood sample at Baseline
* tumor, hemorrhage, aneurysm, hydrocephalus, or other significant clinical finding from Baseline brain MRI

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Regenstrief Institute, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Clark DO, Xu H, Tangney CC, Lin AW, Risacher SL, Saykin AJ, Considine RV, Garringer HJ, Moser L, Carter A, Miller CM, Sprague B, Callahan CM, Unverzagt FW. Feasibility of lifestyle interventions for cognition in adults with low education. Alzheimers Dement. 2025 May;21(5):e70232. doi: 10.1002/alz.70232. PMID 40442881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were excluded from the study before group assignment when Baseline assessment or Tablet Orientation could not be completed.
Period: Immediate Post-Training
Arm/Group | MINDSpeed Intervention | MIND Food and Training Control | Control Foods and Speed of Processing Training | Double Control
Started | 43 | 46 | 45 | 46
Completed | 35 | 44 | 38 | 40
Not Completed | 8 | 2 | 7 | 6
Period: Follow-Up
Arm/Group | MINDSpeed Intervention | MIND Food and Training Control | Control Foods and Speed of Processing Training | Double Control
Started | 35 | 44 | 39 (One participant was active in the study at the end of the Immediate Post-Training period, but did not complete the study visit due to health issues. Participant was still eligible to complete the Follow-Up period, but did not complete the follow-up assessment.) | 40
Completed | 33 | 39 | 38 | 35
Not Completed | 2 | 5 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MINDSpeed Intervention | MIND Food and Training Control | Control Foods and Speed of Processing Training | Double Control | Total
Number analyzed (Participants) | 43 | 46 | 45 | 46 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (6.3) | 65.0 (4.7) | 66.1 (6.4) | 65.6 (5.1) | 65.51 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 28 | 30 | 117
  Male | 12 | 18 | 17 | 16 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 32 | 32 | 30 | 25 | 119
  White | 11 | 12 | 12 | 18 | 53
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 46 | 45 | 46 | 180

OUTCOME MEASURES:

1. Primary Outcome: Executive Cognitive Function Composite Score
Description: Executive Cognitive Function Composite Score as Measured by Individually-Administered Tests of Verbal Fluency, Complex Sequencing, Response Inhibition, and List Learning. The scale score range is -20 to 20. Low scores represent worse function and higher scores represent better function.
Time Frame: Immediately following the 12-week intervention (Immediate Post-Training)]
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MINDSpeed Intervention | MIND Food and Training Control | Control Foods and Speed of Processing Training | Double Control
Number analyzed (Participants) | 43 | 46 | 45 | 46
units on a scale | 0.211 [0.094 to 0.329] | 0.100 [-0.005 to 0.204] | 0.142 [0.029 to 0.254] | 0.196 [0.086 to 0.306]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of study enrollment (i.e., informed consent) until the participant completed the study at 6-Month Follow-Up or withdrew from the study, whichever came first.
Description: Participants were asked specifically about adverse events through structured questionnaire at Immediate Post-Training and Follow-Up study visits, though events were reported throughout the adverse event time frame as they became known to study staff.
Arm/Group | MINDSpeed Intervention | MIND Food and Training Control | Control Foods and Speed of Processing Training | Double Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/46 | 0/45 | 1/46
Serious Adverse Events (participants affected / at risk) | 9/43 | 18/46 | 16/45 | 21/46
Other Adverse Events (participants affected / at risk) | 3/43 | 0/46 | 0/45 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MINDSpeed Intervention (N=43) | MIND Food and Training Control (N=46) | Control Foods and Speed of Processing Training (N=45) | Double Control (N=46)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthma and bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Flu (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mild heart attack (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Assault (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frailty (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Function loss from femur break (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orthopedic surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reactive airway disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toe ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous stasis ulcer (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral illness (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHF complication (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney mass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction rule out (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary track infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Breast cancer (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bunion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cysts (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mobility issues (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nursing home placement (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccine reaction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MINDSpeed Intervention (N=43) | MIND Food and Training Control (N=46) | Control Foods and Speed of Processing Training (N=45) | Double Control (N=46)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03419052/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03419052/ICF_000.pdf